CLINICAL TRIAL: NCT04204057
Title: A Phase 2, Open Label Study to Assess the Efficacy and Safety of Tenalisib (RP6530), a Novel PI3K Dual δ/γ Inhibitor, in Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia (CLL)
Brief Title: Efficacy and Safety of Tenalisib (RP6530) in Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rhizen Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP6530-1901
Record Dates: First submitted 2019-12-04; First posted 2019-12-18 (Actual); Results first posted 2021-07-22 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
Keywords: Phosphoinositide 3-kinase; Pi3k Delta and gamma inhibitor; Tenalisib; Leukemia, Lymphocytic, Chronic, B-Cell
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — tenalisib

STUDY DESIGN:
Intervention Model Description: The trial is a Phase II, open label, Simon's two stage study design to evaluate the efficacy and safety of Tenalisib in patients with CLL who have relapsed or are refractory after at least one prior therapy.
Masking Description: None (open label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tenalisib (Experimental): Patients receive Tenalisib 800 mg BID, Orally in 28-Day cycle for 7 cycles
  Interventions: Drug: Tenalisib

INTERVENTIONS:
Drug: Tenalisib — Tenalisib 800 mg BID, Orally
  Other Names: RP6530

SUMMARY:
The trial is a Phase II, open label, Simon's two stage study design to evaluate the efficacy and safety of Tenalisib in patients with CLL who have relapsed or are refractory after at least one prior therapy.

DETAILED DESCRIPTION:
Tenalisib is a highly specific and orally available dual PI3K δ/γ inhibitor. Pre-clinical experiments demonstrated that Tenalisib is highly effective in killing primary CLL cells in vitro. A Phase II study is planned to evaluate the efficacy and safety of Tenalisib in patients with relapsed/refractory CLL.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosis of B-cell CLL
2. Disease status defined as refractory to or relapsed after at least one prior therapy.
3. Presence of measurable lymphadenopathy presence of > 1 nodal lesion
4. ECOG performance status ≤ 2.
5. Adequate bone marrow, liver, and renal function

Exclusion Criteria:

1. Richter's (large cell) transformation, or PLL transformation.
2. Cancer therapy/ any cancer investigational drug within 3 weeks (21 days) or 5 half-lives (whichever is shorter).
3. Prior exposure to drug that inhibits PI3K
4. Patient with ASCT/Allo-SCT receiving treatment for active GVHD.
5. Ongoing severe systemic bacterial, fungal or viral infection.
6. Central nervous system (CNS) involvement of leukemia or lymphoma.
7. Ongoing immunosuppressive therapy including systemic corticosteroids.
8. Known history of severe liver injury as judge by investigator.
9. Any severe and/or uncontrolled medical conditions or other conditions that could affect patient participation
10. Women who are pregnant or lactating.
11. Known seropositive requiring anti-viral therapy for i. human immunodeficiency virus (HIV) infection. ii. hepatitis B virus (HBV) infection iii. hepatitis c virus (HCV) infection iv. active CMV infection

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Bulgaria (2):
  - University Multiprofile Hospital for Active Treatment "Dr Georgi Stranski" Ltd.,, Pleven
  - University Multiprofile Hospital for Active Treatment "Sv Ivan Rilski" Ltd, Sofia
- Georgia (2):
  - Ltd. M.Zodelava Hematology Centre, Tbilisi
  - Medivest - Institute of Hematology and Transfusiology, Tbilisi
- Poland (2):
  - Silesian Healthy Blood Clinic Grosicki, Grosicka Sp.J., Chorzów
  - Voivodship Multi-Specialist Center for Oncology and Traumatology M. Copernicus, Lodz

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tenalisib
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tenalisib
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 11
Age, Continuous [Median (Full Range); unit: years] | 66.08 [44.93 to 79.27]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Poland | 9
  Georgia | 9
  Bulgaria | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Per Response Evaluation Criteria as defined by iwCLL guideline for CLL: Complete Response (CR), all parameters should be regressed to normal (lymph nodes ≥ 1.5 cm; spleen size <13 cm; liver size normal; no constitutional symptoms; circulating lymphocyte count normal; platelet count ≥ 100 x 109 /L; Hemoglobin ≥ 11.0 g/dL). For partial response, at least two of the parameters (lymph nodes, liver and/or spleen size, constitutional symptoms, circulating lymphocyte count) and one parameter (platelet count, hemoglobin) need to improve if previously abnormal; Overall Response (OR) = CR + PR."
Time Frame: 7 Months
Population: Patients who received at least 1 dose of study medication and provided at least 1 post-baseline efficacy assessment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tenalisib
Number analyzed (Participants) | 21
percentage of participants | 33.3 [14.59 to 56.97]

2. Primary Outcome: Duration of Response (DoR)
Description: Duration of response (DOR): DOR is defined as the interval from the first documentation of CR/PR to the first documentation of definitive disease progression or death from any cause.
  Progression disease is defined using iwCLL criteria as at least one of the criteria of parameters (i.e., lymph nodes increase ≥ 50% from baseline or from response; liver and/or spleen size increase ≥ 50% from baseline or from response; any constitutional symptoms; circulating lymphocyte count increase ≥ 50% over baseline) or criteria of parameters (i.e., platelet count decrease of ≥ 50% over baseline secondary to CLL; hemoglobin decrease of ≥ 50% over baseline secondary to CLL) should be met.
Time Frame: 7 Months
Population: Patients who received at least 1 dose of study medication and provide at least post-baseline efficacy assessment
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Tenalisib
Number analyzed (Participants) | 21
days | 143 [87 to 148]

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events as Assessed by CTCAE Criteria v5.0
Description: Summary of Treatment-Emergent Adverse Events-(Causality All). Patients will be monitored for adverse events and both related and as well as non-related adverse events will be captured during the study. All adverse events (irrespective of causality) will be reported.
Time Frame: 7 Months
Population: Patients who received at least 1 dose of study medication
Measure: Number; unit: participants
Arm/Group | Tenalisib
Number analyzed (Participants) | 21
participants | 15

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival (PFS): PFS is defined as the interval from first dose to first documentation of definitive disease progression or death from any cause.
Time Frame: 7 months
Population: Patients who received at least 1 dose of study medication and provide at least 1 post-baseline efficacy assessment
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Tenalisib
Number analyzed (Participants) | 21
days | 205 [198 to 205]

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Tenalisib
All-Cause Mortality (participants affected / at risk) | 2/21
Serious Adverse Events (participants affected / at risk) | 3/21
Other Adverse Events (participants affected / at risk) | 15/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenalisib (N=21)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenalisib (N=21)
Anemia (Blood and lymphatic system disorders) | 6 (10)
Neutropenia (Blood and lymphatic system disorders) | 5 (18)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 4 (7)
Aspartate aminotransferase increased (Investigations) | 4 (6)
Blood alkaline phosphatase increased (Investigations) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-09-12): https://cdn.clinicaltrials.gov/large-docs/57/NCT04204057/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/57/NCT04204057/SAP_001.pdf